CLINICAL TRIAL: NCT01524549
Title: The Role of the Functionally Relevant Single Nucleotide Polymorphisms CYP2J2 -50G>T (CYP2J2 7) and EPHX2 9846A>G (EPHX2 K55R) in Human Endothelial Function
Brief Title: Blood Vessel Study
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120061; 12-E-0061
Record Dates: First submitted 2012-02-01; First posted 2012-02-02 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-18

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular; P450s; Flow-Mediated Dilation; Brachial Artery Ultrasound; Endothelial Cell Function; Natural History; Healthy Volunteer; HV
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- WT for CYP2J2*7 and heterozygous for EPHX2 K55R: SNP
- WT for CYP2J2*7 and homozygous for EPHX2 K55R: SNP
- WT for EPHX2 K55R and heterozygous for CYP2J2*7: SNP
- WT for EPHX2 K55R and homozygous for CYP2J2*7: SNP
- WT for EPHX2 K55R and WT for CYP2J2*7: SNP

SUMMARY:
Background:

- The endothelium is the inner lining of blood vessels. The cells in this lining help regulate blood flow and immune system function. Problems with endothelial cells can contribute to heart disease, high blood pressure, and diabetes. Certain genes or parts of genes may be related to problems with endothelial function. Researchers want to study healthy adults who have genes that may affect their endothelial function. More information on these genes may provide more information on genetic risk for certain diseases.

Objectives:

- To study healthy adults who have genetic markers related to endothelial cell problems.

Eligibility:

* Healthy volunteers between 18 and 65 years of age.
* Current participants of the Environmental Polymorphisms Registry and have certain genes related to endothelial cell problems.

Design:

* Participants will have a single study visit to collect information and samples.
* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants will have an ultrasound of the artery in the arm and will be given a short-acting medication called nitroglycerin to study blood flow and blood pressure.

DETAILED DESCRIPTION:
According to the CDC, heart disease is the leading cause of death for both men and women of most racial/ethnic groups in the United States, including African Americans, Hispanics, and whites. About 610,000 people die of cardiovascular disease (CVD) every year, accounting for 1 in every 4 deaths (41). Because many known risk factors for heart disease are hereditary, understanding the connection between genetics, particularly heritable polymorphisms, and cardiovascular disease risk is of great importance. This is a cross-sectional, controlled study designed to investigate the association of two single nucleotide polymorphisms (SNPs) - a cytochrome P450 (CYP) epoxygenase gene CYP2J2 SNP, CYP2J2 7, and a soluble epoxide hydrolase (sEH) gene EPHX2 SNP encoding a K55R variant - with altered endothelial function in humans. Healthy adults, aged 18-65 years, who are either carriers of CYP2J2 7 or EPHX2 K55R, or who are wild type (WT) with respect to either SNP will be recruited into a total of five genotype groups. Potential participants will be identified from the Environmental Polymorphisms Registry, mailed an informational letter, contacted by phone and/or email, and pre-screened for eligibility. As participants are recruited, demographic characteristics (i.e., age, gender, and race/ethnicity) will be compared between the groups, and, if necessary, recruitment will be targeted to achieve an approximate match in demographic characteristics across the groups. Pre-screened individuals will provide verbal consent to refrain from taking certain as needed supplements/medications that could alter endothelial function and recreational drugs (such as marijuana, cocaine and amphetamines) prior to the study visit, and will be mailed an informed consent form, medical history form, a urine collection cup, and pre-visit instructions. Participants will attend a single study visit that will take place at the NIEHS Clinical Research Unit. During this visit, written informed consent will be obtained, and there will be a final screening and eligibility determination including medical history review, assessment of vital signs, physical examination, carbon monoxide measurement, pregnancy test (if applicable), and electrocardiogram (ECG). In eligible participants, a lipid panel will be performed and endothelial function will be assessed non-invasively by brachial artery ultrasound (i.e., flow-mediated dilation) and digital peripheral arterial tonometry. Blood and urine (first void) samples will be collected for biomarker analyses, which will be conducted in the Zeldin laboratory at NIEHS. The primary objective of the study is to determine whether individuals who are homozygous or heterozygous for the CYP2J2 7 or EPHX2 K55R SNPs exhibit altered endothelial function compared with individuals who are WT for that SNP. As a secondary objective, the impact of these two SNPs on inflammatory and CYP epoxygenase pathway biomarkers will be examined.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participant of the Environmental Polymorphisms Registry and current contact information available
* Genotype information available for relevant CYP2J2 and EPHX2 polymorphisms, which indicates:

  * WT for EPHX2 K55R and WT for CYP2J2 7
  * WT for EPHX2 K55R and heterozygous for CYP2J2 7
  * WT for EPHX2 K55R and homozygous for CYP2J2 7
  * WT for CYP2J2 7 and heterozygous for EPHX2 K55R (N=30)
  * WT for CYP2J2 7 and homozygous for EPHX2 K55R (N=30)
* Age 18-70 years
* Willing and able to provide informed consent
* Able to comply with all protocol procedures

EXCLUSION CRITERIA:

* Currently pregnant or breast feeding
* Hospitalized for a cardiovascular disease or stroke event within the previous 3 months
* Current use of long-acting nitrates (e.g., isosorbide mononitrate, isosorbide dinitrate)
* Current use of medications taken for hypertension.
* For participants with current daily or chronic use of NSAIDs; unable or unwilling to refrain from taking NSAIDs for 7 days prior to enrollment visit.
* Current use of insulin for Type I Diabetes
* Presence of a pacemaker or implanted cardioverter-defibrillator
* Presence of an irregular heart rhythm (atrial fibrillation) at the study visit
* Current resting heart rate <40 or >125 beats per minute
* Current systolic blood pressure <90 or >180 mmHg, or diastolic blood pressure >110 mmHg
* Skin sensitivity precluding use of ECG electrodes
* History of hypersensitivity to nitroglycerin or other nitrates or nitrites
* History of infection within the preceding 1 week or temperature >38 degrees C
* Unwilling or unable to:

  * Fast (including alcohol and caffeine-containing products) and discontinue tobacco use for 12 hours prior to Visit 1
  * Withhold all prescribed and over-the-counter medications and supplements the morning of Visit 1, until after the visit is completed
  * Refrain from taking the following, as needed, medications for 7 days prior to Visit 1:

    * Vasoactive agents, such as decongestants (e.g., pseudoephedrine)
    * Recreational drugs such as marijuana, cocaine, and amphetamines
    * Anti-inflammatory agents (NSAIDs), such as ibuprofen, naproxen or aspirin
    * Sildenafil (Viagra), vardenafil (Levitra), and tadalafil (Cialis)

Exclusion of Pregnant and Breast Feeding Women: Any woman who is pregnant or breast feeding will be excluded from this study because nitroglycerin, administered as part of the study, is category C, and it is unknown whether nitroglycerin can cause fetal harm when administered to a pregnant woman or whether it can affect reproductive capacity; it is also unknown whether nitroglycerin is excreted in human milk. Also, hormonal changes associated with pregnancy can significantly influence the proposed measures of endothelial function. Females will have a urine pregnancy test prior to undergoing study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Genotype data from the EPR will be used to identify potential study participants@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2012-03-01 (Actual)

PRIMARY OUTCOMES:
-Change in digital pulsatile pressure-Endothelium-independent vasodilation-Change in brachial artery blood flow velocity -Serum levels of inflammatory markers -Serum and urine levels of cytochrome P450 epoxygenase pathway biomarkers@... | analysis
  -Change in digital pulsatile pressure-Endothelium-independent vasodilation-Change in brachial artery blood flow velocity -Serum levels of inflammatory markers -Serum and urine levels of cytochrome P450 epoxygenase pathway biomarkers

SECONDARY OUTCOMES:
-Change in digital pulsatile pressure-Endothelium-independent vasodilation-Change in brachial artery blood flow velocity -Serum levels of inflammatory markers -Serum and urine levels of cytochrome P450 epoxygenase pathway biomarkers@... | analysis
  -Change in digital pulsatile pressure-Endothelium-independent vasodilation-Change in brachial artery blood flow velocity -Serum levels of inflammatory markers -Serum and urine levels of cytochrome P450 epoxygenase pathway biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Darryl C Zeldin, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heron M, Hoyert DL, Murphy SL, Xu J, Kochanek KD, Tejada-Vera B. Deaths: final data for 2006. Natl Vital Stat Rep. 2009 Apr 17;57(14):1-134. PMID 19788058
- [Background] Arking DE, Chakravarti A. Understanding cardiovascular disease through the lens of genome-wide association studies. Trends Genet. 2009 Sep;25(9):387-94. doi: 10.1016/j.tig.2009.07.007. Epub 2009 Aug 26. PMID 19716196
- [Background] Campbell WB, Gebremedhin D, Pratt PF, Harder DR. Identification of epoxyeicosatrienoic acids as endothelium-derived hyperpolarizing factors. Circ Res. 1996 Mar;78(3):415-23. doi: 10.1161/01.res.78.3.415. PMID 8593700
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-E-0061.html